CLINICAL TRIAL: NCT07245693
Title: Longitudinal Assessment of Early Premature Infant Skills for Audiovisual Speech Perception
Acronym: Pré-AV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 38RC24.0246; 2025-A00773-46 (Other: ID/RCB)
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Premature Baby; Neurocognition, Child
Keywords: perception; premature; speech; audiovisual; early skills; nourisson; corrected age; real age; associate; visual speech; auditory speech; language development; aquisition; vocabulary; language difficulties; ASD; capacity; language delay
MeSH Terms: conditions — Premature Birth; Speech; Language Development Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- premature child born before 34 weeks of amenorrhea at the Grenoble Alpes Hospital Center (Experimental): Visits will take place at 4 months of actual age and 4 months of corrected age (i.e., between 6.5-7 months of actual age for a newborn at 28 SA). These appointments will take place within the Neonatology department of the Couple Child Hospital.
  The tests will be carried out by a researcher/student from Babylab, or a pediatric student.
  The measurement of AV association abilities of infants is carried out through comparison of the gaze times of each infant with two speaking faces depending on the sound played in synchrony with the videos. The gaze time with a speaking face congruent with sound compared to the gaze time with a non-congruent speaking face is then coded image by image for each recording of the infant's gaze by 2 independent coders, naive to the hypotheses of the study.
  And one parental questionnaire gathering lists of words usually known and produced by children at term in TTD aged 12 months. It has demonstrated its clinical effectiveness in detecting language delays.
  Interventions: Behavioral: Audiovisual association capability tests

INTERVENTIONS:
Behavioral: Audiovisual association capability tests — Visits will take place at 4 months of actual age and 4 months of corrected age (i.e., between 6.5-7 months of actual age for a newborn at 28 SA). These appointments will take place within the Neonatology department of the Couple Child Hospital. The tests will be carried out by a researcher/student from Babylab, or a pediatric student. The measurement of AV association abilities of infants is carried out through comparison of the gaze times of each infant with two speaking faces depending on the sound played in synchrony with the videos. The gaze time with a speaking face congruent with sound compared to the gaze time with a non-congruent speaking face is then coded image by image for each recording of the infant's gaze by 2 independent coders, naive to the hypotheses of the study. And one parental questionnaire gathering lists of words usually known and produced by children at term in TTD aged 12 months. It has demonstrated its clinical effectiveness in detecting language delays.

SUMMARY:
From birth, babies perceive speech face to face with their interlocutors in audiovisual situations (AV): in addition to hearing them (auditory speech), they will also, in most cases, be able to observe their speaking faces (ex: mouth movements, lips, tongue etc.) . However, the ability to associate visual speech (ex: the movement of the lips of a speaking face) with auditory speech (ex: sound information) to which it corresponds is one of the earliest signs of language development. This ability to audiovisual association is present from the age of 2.5 months in infants with Typical Development and notably allows predicting the subsequent acquisition of vocabulary from the age of 12 months.

This skill allows infants to access redundant AV cues between auditory and visual speech. However this redundancy is a key piece of information allowing them, compared to an auditory situation alone, to focus their attention longer on the speech signal compared to the surrounding noises. This mechanism facilitates their subsequent language learning (identification of sounds, recognition and memorization of vocabulary, etc.) Alternatively, several studies show that children with atypical development of language and communication (e.g., Autistic Spectrum Disorder (ASD)), present clear difficulties in AV association, which may be, at least in part, at the origin of their subsequent linguistic and communicative difficulties.

On the other hand, children born prematurely have a higher risk of language disorders and ASD. Furthermore, some research shows that infants born prematurely exhibit an atypical exploration of speaking faces. This atypicity could explain the subsequent language difficulties observed in these populations.

Currently, we do not know at what age this ability develops in premature children and if it may be the cause of a language development disorder. The hypothesis would be that premature children develop this capacity later than full-term children. This could be one of the explanatory factors for language disorders in the first group. Our study would enrich this AV matching data in premature children and better understand the mechanisms of language delay in them. In addition to other studies, the absence of Matching AV at an expected age could be a strategy for screening for language disorders or ASD in children at risk. This would allow early implementation of intervention programs (speech therapy, parental education...)

ELIGIBILITY:
Inclusion Criteria:

* Born before 34 SA at CHUGA and less than 4 months of actual age
* French mother tongue (i.e., at least one of the two parents is a French mother tongue)
* Legal representatives or parents who have signed a consent to participate in the study.

Exclusion Criteria:

* Severe retinopathies
* Severe neurological damage (grade 3 and 4 intraventricular hemorrhage and periventricular cavity leucomalacia)
* Inconclusive hearing tests

Ages: 4 Months to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion estimated by the ratio of the total gaze time to the speaking face articulating the same sound as that played auditively (congruent) on the total gaze time of the newborn at 4 months of actual age. | From enrollment to the end of treatment at 16 months of life

CONTACTS AND LOCATIONS:
Overall Officials: Marie Dr Chevallier, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: No
confidentiel data

REFERENCES:
- [Background] Imafuku M, Kawai M, Niwa F, Shinya Y, Myowa M. Audiovisual speech perception and language acquisition in preterm infants: A longitudinal study. Early Hum Dev. 2019 Jan;128:93-100. doi: 10.1016/j.earlhumdev.2018.11.001. Epub 2018 Dec 9. PMID 30541680
- [Background] van Noort-van der Spek IL, Franken MC, Weisglas-Kuperus N. Language functions in preterm-born children: a systematic review and meta-analysis. Pediatrics. 2012 Apr;129(4):745-54. doi: 10.1542/peds.2011-1728. Epub 2012 Mar 19. PMID 22430458
- [Background] Arunachalam S, Luyster RJ. The integrity of lexical acquisition mechanisms in autism spectrum disorders: A research review. Autism Res. 2016 Aug;9(8):810-28. doi: 10.1002/aur.1590. Epub 2015 Dec 21. PMID 26688218
- [Background] Irwin JR, Brancazio L. Seeing to hear? Patterns of gaze to speaking faces in children with autism spectrum disorders. Front Psychol. 2014 May 8;5:397. doi: 10.3389/fpsyg.2014.00397. eCollection 2014. PMID 24847297
- [Background] Stevenson RA, Siemann JK, Schneider BC, Eberly HE, Woynaroski TG, Camarata SM, Wallace MT. Multisensory temporal integration in autism spectrum disorders. J Neurosci. 2014 Jan 15;34(3):691-7. doi: 10.1523/JNEUROSCI.3615-13.2014. PMID 24431427
- [Background] Jones W, Klin A. Attention to eyes is present but in decline in 2-6-month-old infants later diagnosed with autism. Nature. 2013 Dec 19;504(7480):427-31. doi: 10.1038/nature12715. Epub 2013 Nov 6. PMID 24196715
- [Background] Weatherhead D, Arredondo MM, Nacar Garcia L, Werker JF. The Role of Audiovisual Speech in Fast-Mapping and Novel Word Retention in Monolingual and Bilingual 24-Month-Olds. Brain Sci. 2021 Jan 16;11(1):114. doi: 10.3390/brainsci11010114. PMID 33467100
- [Background] Newman R, Ratner NB, Jusczyk AM, Jusczyk PW, Dow KA. Infants' early ability to segment the conversational speech signal predicts later language development: a retrospective analysis. Dev Psychol. 2006 Jul;42(4):643-55. doi: 10.1037/0012-1649.42.4.643. PMID 16802897
- [Background] Bahrick LE, Lickliter R. Learning to Attend Selectively: The Dual Role of Intersensory Redundancy. Curr Dir Psychol Sci. 2014 Dec;23(6):414-420. doi: 10.1177/0963721414549187. PMID 25663754
- [Background] Tenenbaum EJ, Sobel DM, Sheinkopf SJ, Shah RJ, Malle BF, Morgan JL. Attention to the mouth and gaze following in infancy predict language development. J Child Lang. 2015 Nov;42(6):1173-90. doi: 10.1017/S0305000914000725. Epub 2014 Nov 18. PMID 25403090
- [Background] Teinonen T, Aslin RN, Alku P, Csibra G. Visual speech contributes to phonetic learning in 6-month-old infants. Cognition. 2008 Sep;108(3):850-5. doi: 10.1016/j.cognition.2008.05.009. Epub 2008 Jun 30. PMID 18590910
- [Background] Birules J, Goupil L, Josse J, Fort M. The Role of Talking Faces in Infant Language Learning: Mind the Gap between Screen-Based Settings and Real-Life Communicative Interactions. Brain Sci. 2023 Aug 5;13(8):1167. doi: 10.3390/brainsci13081167. PMID 37626523
- [Background] Jayaraman S, Smith LB. Faces in early visual environments are persistent not just frequent. Vision Res. 2019 Apr;157:213-221. doi: 10.1016/j.visres.2018.05.005. Epub 2018 Jun 20. PMID 29852210
- See also: French adaptations of short versions of MacArthur-Bates communicative inventories — https://www.researchgate.net/publication/290249718_French_adaptations_of_short_versions_of_MacArthur-Bates_communicative_inventories